CLINICAL TRIAL: NCT03819166
Title: The Effect of Behavioral Support Techniques on Anxiety and Physical Reaction From Dental Treatment
Brief Title: Behavioral Support Techniques on Anxiety and Physical Reaction From Dental Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201012061RC
Record Dates: First submitted 2019-01-14; First posted 2019-01-28 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Dental Anxiety; Dental Diseases; Dental Trauma
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The participants recruited in the group will receive the input of deep touch pressure during their procedures of dental treatment.
  Interventions: Device: with deep touch pressure application
- control group (Sham Comparator): The participants recruited in the group will not receive the input of deep touch pressure during their procedures of dental treatment.
  Interventions: Device: without deep touch pressure application

INTERVENTIONS:
Device: with deep touch pressure application — The deep touch pressure is applied by the weight loading devices, including but not limited to, weight blanket and weight vest.
  Arms: experimental group
Device: without deep touch pressure application — The deep touch pressure will not be applied.
  Arms: control group

SUMMARY:
Application of deep touch pressure (DTP) has been suggested to provide positive effects on anxiety modulation. However, empirical and theoretical evidence linked to the clinical effects of DTP is relatively rare in the behavioral and physiological aspects. The aim of this intervention trial study designs to investigate the effect of DTP in dental treatment by quantitative analysis of behavioral assessments and physiological measurements, including the electrodermal activity and heart rate variability, were conducted to understand the modulation of the autonomic nervous system (ANS), the orchestration of sympathetic (SNS) and parasympathetic (PsNS) nervous systems.

DETAILED DESCRIPTION:
The subjects were recruited through word-of-mouth and by posted sign-up from the Department of Dentistry, National Taiwan University Hospital (NTUH), Taiwan. Informed consent was obtained prior to participation. The study protocol was approved by the Human Research Ethics Committee of NTUH. Before the testing, the experimental protocol was explained to the subjects. The subjects with normal overnight sleep quality were recruited to prevent the influences in both physiological and physical fatigue. All potential subjects receive independent examinations by an occupational therapist and a dentist to determine the eligibility for inclusion as well as were blind to the study hypotheses. Both electrodermal activity (EDA) and heart rate variability (HRV) were recorded continually through the entire testing procedures. Since the EDA and HRV are sensitive indicators for autonomic nervous system modulation, a standardization procedure that ensures the integrity of data is accessed. The power of the testing is preset at 0.80, and the significant level is 0.05. The quasi-experimental design of clinical trial for repeated measures will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients who requiring tooth extraction were potentially selected to recruit.

Exclusion Criteria:

* with a history of systemic diseases that would contraindicate surgical treatment
* pregnant and lactating
* smoking of more than 10 cigarettes per day
* poor overnight sleep quality
* refusal to sign the inform consent agreement

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03-11 (Actual); Primary Completion 2013-07-18 (Actual); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability (HRV) | The baseline phase is defined as the five minutes before the dental treatment. The HRV data recorded in this phase will be considered as the baseline data of this study.
  A non-invasive technique to investigate the effect of mental stress of the autonomic nervous system control on heart rate.
Electrodermal Activity (EDA) | The baseline phase is defined as the five minutes before the dental treatment. The EAD data recorded in this phase will be considered as the baseline data of this study
  A non-invasive technique to investigate the effect of mental stress of the sympathetic nervous system control on sweat gland of skin.
Heart Rate Variability (HRV) | The treatment phase is the period of the entire procedures of dental treatment, approximate 40-90 minutes. The HRV data will be recorded to investigate the changes both during the dental treatment and in the application of deep touch pressure.
  A non-invasive technique to investigate the effect of mental stress of the autonomic nervous system control on heart rate.
Electrodermal Activity (EDA) | The treatment phase is the period of the entire procedures of dental treatment, approximate 40-90 minutes. The EDA data will be recorded to investigate the changes both during the dental treatment and in the application of deep touch pressure.
  A non-invasive technique to investigate the effect of mental stress of the sympathetic nervous system control on sweat gland of skin.
Heart Rate Variability (HRV) | The post-treatment phase is defined as the five minutes after the dental treatment. The HRV data recorded in this phase will be considered as the post-treatment data which used to compare to the baseline and treatment data.
  A non-invasive technique to investigate the effect of mental stress of the autonomic nervous system control on heart rate.
Electrodermal Activity (EDA) | The post-treatment phase is defined as the five minutes after the dental treatment. The EDA data recorded in this phase will be considered as the post-treatment data which used to compare to the baseline and treatment data.
  A non-invasive technique to investigate the effect of mental stress of the sympathetic nervous system control on sweat gland of skin.

SECONDARY OUTCOMES:
Dental Anxiety Scale (DAS) | This questionnaire will be applied in the baseline phase (immediately after HRV measurement and about 5 minutes before dental procedures) to know anxiety condition of participants before the dental treatment.
  This questionnaire can range from 4 (not anxious at all) to 20 (extremely anxious).
Dental Anxiety Scale (DAS) | The averaged time of dental treatment is about 40-90 minutes.This questionnaire will be applied immediately after the dental treatment completion.
  This questionnaire can range from 4 (not anxious at all) to 20 (extremely anxious).
Numeric State Anxiety Scale (NSAS) | This scale will be scored in the baseline phase (immediately after HRV measurement and about 5 minutes before dental procedures) to identify the anxiety state of participants before the dental treatment.
  This ordinal scale, range from 0-10, which is represented as a abscissa line to reflect the level of anxiety; 0 and 1 is not at all, 2 to 4 is little, 5 to 7 is medium, 8 and 9 is a lot, and 10 is worst imaginable.
Numeric State Anxiety Scale (NSAS) | The averaged time of dental treatment is about 40-90 minutes.This scale will be scored immediately after the dental treatment completion.
  This ordinal scale, range from 0-10, which is represented as a abscissa line to reflect the level of anxiety; 0 and 1 is not at all, 2 to 4 is little, 5 to 7 is medium, 8 and 9 is a lot, and 10 is worst imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiagn Yang, DDS, Principal Investigator — Department of Dentistry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.